CLINICAL TRIAL: NCT03397407
Title: Lifestyle, Adiposity, and Cardiovascular Health in Youth Study
Brief Title: Lifestyle, Adiposity, and Cardiovascular Health in Youth
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Other Study IDs: AugustaU
Record Dates: First submitted 2017-12-18; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Lifestyle; Adiposity; Cardiovascular Diseases; Adolescent
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Adiposity is a key link between lifestyle factors (like diet and exercise) and cardiovascular (CV) disease. However, little is known about the link during the juvenile years, when the processes leading to CV disease are at an early stage of development. The specific aims are as follow: (1) to determine the relations of free-living diet and exercise to total body percent fat ( percentBF), visceral adipose tissue and CV fitness in black and white boys and girls of varying socioeconomic status. (2) to determine the relations of fatness and fitness to different CV disease risk factors. Design and methods: (1) Recruit 800 14 to 18 year olds, 200 in each ethnicity and gender subgroup. (2) Assess diet with seven 24-hour recalls, and exercise with two seven-day recalls and heart rate monitoring. (3) Measure percent body fat with dual-energy x-ray absorptiometry, visceral adipose tissue with magnetic resonance imaging and CV fitness with a multi-stage treadmill test. (4) Measure major fatness- and fitness-related CV disease risk factors (e.g., total cholesterol:HDL cholesterol ratio, insulin, systolic blood pressure, left ventricular mass indexed to height, fibrinogen). (5) Conduct multivariate and univariate analyses to determine relationships.

DETAILED DESCRIPTION:
Adult studies have shown that adiposity, especially visceral adipose tissue, and cardiovascular (CV) fitness are key links between lifestyle factors like diet and exercise on one hand, and CV disease on the other. However, very little is known about these links during the juvenile years, when the processes leading to CV disease are at an early stage of development. The specific aims are as follow: (1) to determine the relations of free-living diet and exercise to total body percent fat ( percent BF), visceral adipose tissue and CV fitness in black and white boys and girls of varying socioeconomic status. (2) to determine the relations of fatness and fitness to different CV risk factors. Design and methods: (1) Recruit 800 14 to 18 year olds, 200 in each ethnicity and gender subgroup. (2) Assess diet with seven 24-hour recalls, and exercise with two seven-day recalls and Actigraph monitors. (3) Measure percent body fat with dual-energy x-ray absorptiometry, visceral adipose tissue with magnetic resonance imaging and CV fitness with a multi-stage treadmill test. (4) Measure major fatness- and fitness-related CV disease risk factors (e.g., total cholesterol:HDL cholesterol ratio, insulin, systolic blood pressure, left ventricular mass indexed to height, fibrinogen). (5) Conduct multivariate and univariate analyses to determine relationships. Health relatedness: The provided by this project will assist in the formulation of effective lifestyle interventions targeted to specific demographic groups for primary prevention of CV disease, starting early in life when the foundations for adult disease are being laid.

ELIGIBILITY:
Inclusion Criteria:

* European or African American and age 14-18 years

Exclusion Criteria:

* Taking medications or had any chronic medical conditions that might affect growth, maturation, physical activity, nutritional status, or metabolism.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Recruit 800 14 to 18 year olds, 200 in each ethnicity (European or African American) and gender subgroup.
Sampling Method: Non-Probability Sample
Enrollment: 796 (Actual)
Dates: Start 2001-08-01 (Actual); Primary Completion 2004-07-31 (Actual); Study Completion 2005-01-01 (Actual)

PRIMARY OUTCOMES:
Fatness | Through study completion, an average of 4 years
  Percentage of body fat (%)
Fitness | Through study completion, an average of 4 years
  Maximal oxygen consumption (VO2, mL/kg/min)
Insulin resistance | Through study completion, an average of 4 years
  Fasting insulin (pmol/L)

SECONDARY OUTCOMES:
Fat distribution | Through study completion, an average of 4 years
  Visceral adipose tissue volume (cm^3)
Cardiovascular risk factor | Through study completion, an average of 4 years
  Triglyceride (TG, mmol/L) and high density lipoprotein cholesterol (HDLC, mmol/L) will be combined to report TG/HDLC ratio